CLINICAL TRIAL: NCT02939638
Title: A Randomized, Controlled Trial on Diet, Insulin Sensitivity, and Postprandial Metabolism
Brief Title: Diet, Insulin Sensitivity, and Postprandial Metabolism
Acronym: TEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00018983
Record Dates: First submitted 2016-10-17; First posted 2016-10-20 (Estimated); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Overweight; Obesity; Insulin Resistance
Keywords: Plant-based diet; Obesity; Insulin sensitivity; Intracellular lipid; Postprandial metabolism; Vegan diet; Beta-cell function
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance | interventions — Diet, Plant-Based; Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plant-based diet (Active Comparator): The diet group will be asked to follow a low-fat, vegan diet for 16 weeks
  Interventions: Other: Plant-based diet
- Control diet (Active Comparator): Half of the participants will be asked to continue their usual diets for the 16-week study period.
  Interventions: Other: Control Diet

INTERVENTIONS:
Other: Plant-based diet — Weekly instructions will be given to the participants in the intervention group about following vegan diet.
  Other Names: Vegan diet
  Arms: Plant-based diet
Other: Control Diet — Participants will be asked to continue their usual diets for the 16-week study period.
  Arms: Control diet

SUMMARY:
This randomized, controlled trial aims to elucidate the mechanisms by which a plant-based dietary intervention causes weight loss. Using a low-fat, plant-based diet for 16 weeks, along with an untreated control for comparison, the study will measure changes in body weight, body composition, intramyocellular and/or intrahepatocellular lipid, and changes in association to body weight.

DETAILED DESCRIPTION:
In a 16-week trial, overweight adults will be randomly assigned to two groups. Changes in body weight, body composition, intramyocellular and/or intrahepatocellular lipid, and changes in association to body weight will be measured among other outcomes.

The Intervention Group will follow a low-fat, vegan diet and will receive weekly classes and support.

The Control Group will be asked to follow a conventional control diet.

This study conducts a pilot sub-study to test the hypothesis that changes in insulin sensitivity and beta-cell function observed in response to a diet intervention correlate with changes in intramyocellular and/or intrahepatocellular lipid. Another sub-study assesses the association between metabolic outcomes and gut microbiome. One additional sub-study is looking for associations between metabolic outcomes and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age ≥18 years of age
* Body mass index 28-40 kg/m2

Exclusion Criteria:

1. Diabetes mellitus, type 1 or 2, history of diabetes mellitus or of any endocrine condition that would affect body weight, such as thyroid disease, pituitary abnormality, or Cushing's syndrome
2. Smoking during the past six months
3. Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
4. Use of recreational drugs in the past 6 months
5. Use within the preceding six months of medications that affect appetite or body weight, such as estrogens or other hormones, thyroid medications, systemic steroids, antidepressants (tricyclics, monoamine oxidase inhibitors (MAOIs), selective serotonin reuptake inhibitors (SSRIs), antipsychotics, lithium, anticonvulsants, appetite suppressants or other weight-loss drugs, herbs for weight loss or mood, St. John's wort, ephedra, beta blockers
6. Pregnancy or intention to become pregnant during the study period
7. Unstable medical or psychiatric illness
8. Evidence of an eating disorder
9. Likely to be disruptive in group sessions
10. Already following a low-fat, vegan diet
11. Lack of English fluency
12. Inability to maintain current medication regimen
13. Inability or unwillingness to participate in all components of the study
14. Intention to follow another weight-loss method during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Body weight in kg | 16 weeks
  Anticipated weight-loss for intervention group compared with control group. Weight and height will be combined to report BMI in kg/m^2
Fat mass in grams | 16 weeks
  Anticipated weight-loss for intervention group compared with control group.
Visceral fat in cm^3 | 16 weeks
  Anticipated weight-loss for intervention group compared with control group.
Changes in intramyocellular and/or intrahepatocellular lipid | 16 Weeks
  A subset of participants will be selected for magnetic resonance (MR) spectroscopy studies quantifying hepatic lipid and/or intramyocellular and/or contents in order to provide data regarding possible causal relationships between dietary changes, ectopic lipid, and insulin sensitivity. Selected individuals with varying degrees of insulin-resistance in both groups will be assessed before and after the intervention period. These magnetic resonance spectroscopy (MRS) studies will take place at the Magnetic Research Center at Yale University School of Medicine, New Haven, CT.
Insulin resistance | 16 weeks
  Insulin resistance will be assessed by the Homeostatic Model Assessment (HOMA) index.
Resting Energy Expenditure (REE) | 16 weeks
  Participants will be asked to report to the laboratory within 60 minutes of waking and after a 12-hour fast. Following 30 minutes of quiet rest in a dimly lit room, pulse, respiratory rate, and body temperature will be measured. REE will be measured for 20 minutes through indirect calorimetry (COSMED Metabolic Company Quark Resting Metabolic Rate (RMR), Chicago, IL) utilizing a ventilated hood system. The laboratory temperature will be maintained at 23 degrees C throughout, and precautions will be taken to minimize any disturbances that could affect the metabolic rate. For premenopausal women, measures will be timed so as to occur in the luteal phase of the menstrual cycle.
Postprandial metabolism | 16 weeks
  Participants will be asked to report to the laboratory within 60 minutes of waking and after a 12-hour fast. Postprandial metabolism will be measured for three hours after the standard meal. For premenopausal women, measures will be timed so as to occur in the luteal phase of the menstrual cycle.

SECONDARY OUTCOMES:
Beta-cell function as measured by glucose (mmmol/L) | 16 weeks
  A standard meal test will be performed after an overnight fast. Plasma glucose, will be measured at 0, 30, 60, 120, and 180 min for a total of 3-hours over a 16-week period. Glucose, insulin and C-peptide will combined and analyzed to report Beta-cell function.
Beta-cell function as measured by insulin (pmol/L) | 16 weeks
  A standard meal test will be performed after an overnight fast. Plasma insulin will be measured at 0, 30, 60, 120, and 180 min for a total of 3-hours over a 16-week period. Glucose, insulin and C-peptide will combined and analyzed to report Beta-cell function.
Beta-cell function as measured by C-peptide (ng/mL) | 16 weeks
  A standard meal test will be performed after an overnight fast. Plasma C-peptide will be measured at 0, 30, 60, 120, and 180 min for a total of 3-hours over a 16-week period. Glucose, insulin and C-peptide will combined and analyzed to report Beta-cell function.
Microbiome Analysis | 16 weeks
  Microbiome analysis from participant-provided stool sample. Analysis from uBiome Biotechnology company in a subset of participants. Anticipated changes in the dietary intervention group include changes in the microbiome composition that correlate with changes in insulin sensitivity.
Endothelial function | 16 weeks
  Endothelial function will be measured using the EndoPAT, a proprietary diagnostic device for functional vascular health assessment, in a subset of participants.
Diet Assessment Recall Questionnaire | 16 weeks
  24-hour multi-pass dietary recalls will be used to assess dietary adherence to assist study personnel in working with individuals who need additional teaching or support.
The Effect of Fat Quantity & Quality on Body Composition, Insulin Resistance, & Insulin Secretion | 16 Weeks
  Regression Analysis will be used to assess The Effect of Fat Quantity & Quality on Body Composition, Insulin Resistance, & Insulin Secretion
The Effect of Carbohydrate Quantity & Quality on Body Composition & Insulin Resistance | 16 Weeks
  Regression Analysis will be used to assess The Effect of Carbohydrate Quantity & Quality on Body Composition & Insulin Resistance
The Effect of Protein Quantity & Quality on Body Composition, Insulin Resistance, & Insulin Secretion | 16 Weeks
  Regression Analysis will be used to assess The Effect of Protein Quantity & Quality on Body Composition, Insulin Resistance, & Insulin Secretion
Levels of Advanced Glycosylation Endproducts (AGEs) | 16 Weeks
  An AGE reader will be used to measure the Levels of the AGEs in the skin
Race Disparities | 16 weeks
  Compare the effectiveness of the vegan diet in Blacks vs. Whites in all the primary outcomes
Dietary Advanced Glycation End Products (AGEs) | 16 weeks
  Explore the effectiveness of a vegan diet in reducing dietary AGEs.
Food costs | 16 weeks
  Food costs will be assessed, using the U.S. Department of Agriculture Thrifty Food Plan, 2021, at baseline and 16 weeks.
PDI, hPDI, uPDI | 16 weeks
  Assess the total plant-based index (PDI), healthy PDI, and unhealthy PDI, and their relationship with weight loss
Ultraprocessed foods | 16 weeks
  The consumption of ultraprocessed foods will be assessed, using the NOVA classification, at baseline and 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Neal D Barnard, M.D., Principal Investigator — President
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tonstad S, Butler T, Yan R, Fraser GE. Type of vegetarian diet, body weight, and prevalence of type 2 diabetes. Diabetes Care. 2009 May;32(5):791-6. doi: 10.2337/dc08-1886. Epub 2009 Apr 7. PMID 19351712
- [Background] Barnard ND, Levin SM, Yokoyama Y. A systematic review and meta-analysis of changes in body weight in clinical trials of vegetarian diets. J Acad Nutr Diet. 2015 Jun;115(6):954-69. doi: 10.1016/j.jand.2014.11.016. Epub 2015 Jan 22. PMID 25620754
- [Background] Barnard ND, Scialli AR, Turner-McGrievy G, Lanou AJ, Glass J. The effects of a low-fat, plant-based dietary intervention on body weight, metabolism, and insulin sensitivity. Am J Med. 2005 Sep;118(9):991-7. doi: 10.1016/j.amjmed.2005.03.039. PMID 16164885
- [Background] Shulman GI. Ectopic fat in insulin resistance, dyslipidemia, and cardiometabolic disease. N Engl J Med. 2014 Sep 18;371(12):1131-41. doi: 10.1056/NEJMra1011035. No abstract available. PMID 25229917
- [Background] Petersen KF, Dufour S, Morino K, Yoo PS, Cline GW, Shulman GI. Reversal of muscle insulin resistance by weight reduction in young, lean, insulin-resistant offspring of parents with type 2 diabetes. Proc Natl Acad Sci U S A. 2012 May 22;109(21):8236-40. doi: 10.1073/pnas.1205675109. Epub 2012 Apr 30. PMID 22547801
- [Background] Sparks LM, Xie H, Koza RA, Mynatt R, Hulver MW, Bray GA, Smith SR. A high-fat diet coordinately downregulates genes required for mitochondrial oxidative phosphorylation in skeletal muscle. Diabetes. 2005 Jul;54(7):1926-33. doi: 10.2337/diabetes.54.7.1926. PMID 15983191
- [Background] Goff LM, Bell JD, So PW, Dornhorst A, Frost GS. Veganism and its relationship with insulin resistance and intramyocellular lipid. Eur J Clin Nutr. 2005 Feb;59(2):291-8. doi: 10.1038/sj.ejcn.1602076. PMID 15523486
- [Background] Barnard ND, Gloede L, Cohen J, Jenkins DJ, Turner-McGrievy G, Green AA, Ferdowsian H. A low-fat vegan diet elicits greater macronutrient changes, but is comparable in adherence and acceptability, compared with a more conventional diabetes diet among individuals with type 2 diabetes. J Am Diet Assoc. 2009 Feb;109(2):263-72. doi: 10.1016/j.jada.2008.10.049. PMID 19167953
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Petersen KF, Dufour S, Feng J, Befroy D, Dziura J, Dalla Man C, Cobelli C, Shulman GI. Increased prevalence of insulin resistance and nonalcoholic fatty liver disease in Asian-Indian men. Proc Natl Acad Sci U S A. 2006 Nov 28;103(48):18273-7. doi: 10.1073/pnas.0608537103. Epub 2006 Nov 17. PMID 17114290
- [Background] Gruetter R. Automatic, localized in vivo adjustment of all first- and second-order shim coils. Magn Reson Med. 1993 Jun;29(6):804-11. doi: 10.1002/mrm.1910290613. PMID 8350724
- [Background] Rabol R, Petersen KF, Dufour S, Flannery C, Shulman GI. Reversal of muscle insulin resistance with exercise reduces postprandial hepatic de novo lipogenesis in insulin resistant individuals. Proc Natl Acad Sci U S A. 2011 Aug 16;108(33):13705-9. doi: 10.1073/pnas.1110105108. Epub 2011 Aug 1. PMID 21808028
- [Background] American Dietetic Association; Dietitians of Canada. Position of the American Dietetic Association and Dietitians of Canada: Vegetarian diets. J Am Diet Assoc. 2003 Jun;103(6):748-65. doi: 10.1053/jada.2003.50142. PMID 12778049
- [Background] Barnard ND, Akhtar A, Nicholson A. Factors that facilitate compliance to lower fat intake. Arch Fam Med. 1995 Feb;4(2):153-8. doi: 10.1001/archfami.4.2.153. PMID 7842153
- [Background] Buzzard IM, Faucett CL, Jeffery RW, McBane L, McGovern P, Baxter JS, Shapiro AC, Blackburn GL, Chlebowski RT, Elashoff RM, Wynder EL. Monitoring dietary change in a low-fat diet intervention study: advantages of using 24-hour dietary recalls vs food records. J Am Diet Assoc. 1996 Jun;96(6):574-9. doi: 10.1016/S0002-8223(96)00158-7. PMID 8655904
- [Derived] Kahleova H, Brennan H, Znayenko-Miller T, Holubkov R, Barnard ND. Does diet quality matter? A secondary analysis of a randomized clinical trial. Eur J Clin Nutr. 2024 Mar;78(3):270-273. doi: 10.1038/s41430-023-01371-y. Epub 2023 Nov 28. PMID 38012413
- [Derived] Kahleova H, Sutton M, Maracine C, Nichols D, Monsivais P, Holubkov R, Barnard ND. Vegan Diet and Food Costs Among Adults With Overweight: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2332106. doi: 10.1001/jamanetworkopen.2023.32106. PMID 37669055
- [Derived] Kahleova H, Znayenko-Miller T, Uribarri J, Holubkov R, Barnard ND. Dietary advanced glycation products and their associations with insulin sensitivity and body weight: A 16-week randomized clinical trial. Obes Sci Pract. 2022 Oct 21;9(3):235-242. doi: 10.1002/osp4.646. eCollection 2023 Jun. PMID 37287522
- [Derived] Kahleova H, Rembert E, Nowak A, Holubkov R, Barnard ND. Effect of a diet intervention on cardiometabolic outcomes: Does race matter? A randomized clinical trial. Clin Nutr ESPEN. 2021 Feb;41:126-128. doi: 10.1016/j.clnesp.2020.12.012. Epub 2021 Jan 2. PMID 33487254
- [Derived] Kahleova H, Petersen KF, Shulman GI, Alwarith J, Rembert E, Tura A, Hill M, Holubkov R, Barnard ND. Effect of a Low-Fat Vegan Diet on Body Weight, Insulin Sensitivity, Postprandial Metabolism, and Intramyocellular and Hepatocellular Lipid Levels in Overweight Adults: A Randomized Clinical Trial. JAMA Netw Open. 2020 Nov 2;3(11):e2025454. doi: 10.1001/jamanetworkopen.2020.25454. PMID 33252690